CLINICAL TRIAL: NCT05706077
Title: Effects of tDCS and Physical Therapy on Pain in Women With Chronic Migraine: A Factorial Clinical Trial Randomized, Blinded
Brief Title: Effects of tDCS and Physical Therapy in Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Renata Emanuela Lyra de Brito Aranha, principal investigator, master's degree in cognitive and behavioral neuroscience, Federal University of Paraíba
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 65756722.6.0000.5188
Record Dates: First submitted 2022-12-29; First posted 2023-01-31 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Migraine Disorders
Keywords: physical therapy; transcranial direct current stimulation; facial recognition
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into four intervention groups: transcranial Direct Current Stimulation + Physical Therapy Group (tDCS active + PT active), tDCS group (tDCS active + PT placebo), PT group (tDCS sham + PT active), control group (tDCS sham + PT placebo ).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- active tDCS + real Physical Therapy (Experimental): Active Transcranial Direct Current Stimulation will be applied associated with real physiotherapy. The electrode position will be performed according to the 10-20 international system of marking and the different montages will be realized by distinct application sites.
  To stimulate the primary motor cortex the active electrode will be positioned on the C3 point and the reference electrode on the contralateral supraorbital region.
  Interventions: Device: active tDCS; Other: real Physical Therapy
- active tDCS + placebo Physical Therapy (Placebo Comparator): Active Transcranial Direct Current Stimulation will be applied associated with placebo physiotherapy. The electrode position will be performed according to the 10-20 international system of marking and the different montages will be realized by distinct application sites.
  To stimulate the primary motor cortex the active electrode will be positioned on the C3 point and the reference electrode on the contralateral supraorbital region.
  Interventions: Device: active tDCS; Other: placebo Physical Therapy
- sham tDCS + real Physical Therapy (Sham Comparator): Sham Transcranial Direct Current Stimulation will be applied associated with real physiotherapy. The electrode position will be performed according to the 10-20 international system of marking and the different montages will be realized by distinct application sites. The anode electrode will be positioned on the C3 point (primary motor cortex) and the reference electrode on the contralateral supraorbital region.
  Interventions: Device: sham tDCS; Other: real Physical Therapy
- sham tDCS + placebo Physical Therapy (Other): Sham Transcranial Direct Current Stimulation will be applied associated with placebo physiotherapy. The electrode position will be performed according to the 10-20 international system of marking and the different montages will be realized by distinct application sites. The anode electrode will be positioned on the C3 point (primary motor cortex) and the reference electrode on the contralateral supraorbital region.
  Interventions: Device: sham tDCS; Other: placebo Physical Therapy

INTERVENTIONS:
Device: active tDCS — The electrode will measure 5x5 cm and a current of 2mA will be applied for 20 minutes. The current density will be 0.08mA/cm². tDCS will be applied three times a week for 20 minutes over four weeks.
  Arms: active tDCS + placebo Physical Therapy; active tDCS + real Physical Therapy
Device: sham tDCS — The electrode will measure 5x5 cm. The sham-type current will show a rising ramp where the initial 30 seconds will be real current with the same parameter as the active group. After this time, the current will be automatically stopped by the device. tDCS will be applied three times a week for 20 minutes over four weeks.
  Arms: sham tDCS + placebo Physical Therapy; sham tDCS + real Physical Therapy
Other: real Physical Therapy — Manual maneuvers and therapeutic exercises will be performed for 30 minutes, three times a week over four weeks.
  Arms: active tDCS + real Physical Therapy; sham tDCS + real Physical Therapy
Other: placebo Physical Therapy — The placebo Physical Therapy will be applied for 30 minutes, three times a week over four weeks. The initial 20 minutes will be used for the application of simulated ultrasound bilaterally in the middle portion of the upper trapezius muscle. In the final 10 minutes, the researcher will place the palms of the hand under the occipital region without applying any force or movement with the participant in the supine position.
  Arms: active tDCS + placebo Physical Therapy; sham tDCS + placebo Physical Therapy

SUMMARY:
The aim of this clinical study is to compare the effects of tDCS, physiotherapy, and their association with the intensity in women with Chronic Migraine. For this purpose, the patients included in the study will be distributed among four groups following a factorial model.

DETAILED DESCRIPTION:
A factorial, randomized clinical trial will be conducted to evaluate pain control, the number of migraine attacks, quality of life, emotional dysfunctions, and attentional processing of migraine patients.

Clinical outcomes will be evaluated through (I) a Visual Analog Scale (VAS); (II) pressure pain threshold; (III) a Headache Impact Test (HIT-6); (IV) a Migraine Disability Assessment (MIDAS); (V) Short-Form Health Survey Questionnaire de 36 items (SF-36); (VI) Patients' Global Impression of Change Scale (PGICS); (VII) Beck Depression Inventory (BDI); (VIII) State-Trait Anxiety Inventory (S-TAI); (IX) Perceived Stress Scale (PSS); and (X) Facial Expression Database.

ELIGIBILITY:
Inclusion Criteria:

* Women;
* 18-50 years old;
* with Chronic Migraine according to ICHD-3 beta;
* literate;
* stable on routine medications specific for MC for at least 2 months, who were not undergoing other types of non-pharmacological interventions for MC, not lactating or pregnant, without neurological diseases or serious neuropsychiatric diseases, without other types of associated headaches, without signs and/or symptoms of spinal radiculopathy, without metal implants located in the head and/or cochlear implants.

Exclusion Criteria:

* who perhaps become pregnant during the execution of the clinical trial
* present some disease that disables their continuity in the treatment
* start another type of treatment
* show changes in physical activity and/or eating routine during the research
* has severe depression (BDI > 35).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2023-03-25 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Visual Analogic Scale | baseline, one month, two month
  This scale will be used to measure the patients' pain intensity. The scale consists of a 100 mm line within the limits of no pain and worst possible pain. The patient is instructed to trace the intensity of his pain within the limits of the line. Changes of 1.1 to 1.2 cm indicate minimal clinical improvement.
pressure pain threshold | baseline, one month, two month
  We analyzed the following points with the pressure algometer: anterior and posterior fibers of the temporal muscle, frontal region, insertion of the sternocleidomastoid muscle, insertion and middle fibers of the upper trapezius muscle, thenar region of the right upper limb.

SECONDARY OUTCOMES:
Headache Impact Test | baseline, one month, two month
  This test assesses the impact of headache on quality of life. A total score less than 50 means no severity; between 50 and 55, some severity; between 56 and 59, substantial severity; greater than 60, severe impact.
Migraine Disability Assessment | baseline, one month, two month
  This questionnaire assesses the inability to perform activities of daily living of people with migraine.The MIDAS score is divided into grades: Grade I - little or no disability (scores 0-5), grade II - mild disability (scores 6-10), grade III - moderate disability (scores 11-20), and grade IV - severe disability (score equal to or greater than 21).
Short-Form Health Survey Questionnaire | baseline, one month, two month
  This questionnaire assesses health-related quality of life. This test consists of 36 items. Higher scores indicate greater functionality.
Patients' Global Impression of Change Scale | baseline, one month, two month
  This scale rates the improvement associated with the intervention on a 7-item scale ranging from "1=no change" to "7=much better".
Beck Depression Inventory | baseline, one month, two month
  This questionnaire assesses the participants' level of depression. Scores between 0-11 mean minimal depression; between 12-19: mild depression; between 20-35: moderate depression and between 36-63: severe depression.
State-Trait Anxiety Inventory | baseline, one month, two month
  This instrument assesses the participants' anxiety. It consists of 40 statements that consider trait anxiety and state anxiety. Answers are given on a four-point Likert-type scale (1 - not to 4 - very much), and the score can vary between 20-80. Anxiety level classification can be low (20-33 points), medium (33-49 points), and high (49-80 points).
Perceived Stress Scale | baseline, one month, two month
  It is an instrument composed of 14 questions with response options ranging from zero to four (0=never; 1=almost never; 2=sometimes; 3=almost always, and 4=always). Questions with a positive connotation (4, 5, 6, 7, 9, 10, and 13) have their scores inverted: 0=4, 1=3, 2=2, 3=1, and 4=0. The other questions have negative valence and are added directly. The score is the sum of the scores for each question and can range from 0 to 56.
Facial Expression Database | baseline, one month, two month
  This is an instrument that evaluates the recognition of facial expressions. The bank of faces from Lacop - Facial Expression Database will be used with expressions of joy, fear, anger, sadness, disgust, and surprise from two male and two female models. The manipulation of the intensity of the expressions will be carried out through the Morpheus 4.0 Software to generate faces with different emotional intensities with incremental advances of 25% from the neutral face until reaching 100% of expression intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Renata Aranha, Principal Investigator — Federal University of Paraiba
Locations (1):
- Federal University of Paraiba, João Pessoa, Paraíba, Brazil